CLINICAL TRIAL: NCT06888141
Title: Virtual Intervention Targeting Distress in College Students: A Pilot Study
Brief Title: Stress Management for College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Matt Genuchi, Associate Professor, Boise State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB24-765; U01GM152530 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Distress, Emotional
Keywords: virtual intervention; men/male; college students; emotional distress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Intervention (Experimental)
  Interventions: Behavioral: Virtual Sequential Emotional Processing Task
- Virtual Control (Sham Comparator)
  Interventions: Behavioral: Virtual Control Task

INTERVENTIONS:
Behavioral: Virtual Sequential Emotional Processing Task — A 20-minute interactive session delivered 3 times over a one week period.
  Arms: Virtual Intervention
Behavioral: Virtual Control Task — A time-matched (ie., 20 minute) interactive session delivered 3 times over a one week period.
  Arms: Virtual Control

SUMMARY:
The goal of this clinical trial is to learn if a virtual task can reduce distress in college students. The main questions it aims to answer are:

1. Will those who complete the virtual task have less distress?
2. Will men and women both benefit equally from the virtual task?

Researchers will compare the virtual task to a control task (another virtual task that we expect will not impact distress) to see if distress differs.

Participants will spend 20 minutes engaging in the virtual task (or the control task) on 3 different days all within one week. They will complete a survey about their well-being before starting the first virtual task and again ~6 weeks afterward.

DETAILED DESCRIPTION:
Easily accessible and cost effective strategies for reducing emotional distress and improving stress tolerance in college students and the population generally are desired. The scalability and feasibility of virtual interventions hold promise for reaching segments of the population that find one-on-one psychotherapy aversive. Males in particular have higher perceived treatment stigma relative to women and find may typical traditional therapeutic processes incongruent with their masculine identity and values. The research team has designed an innovative, self-directed, virtual intervention to reduce distress and stress intolerance. The intervention consists of a set of virtual tasks which reflect the Sequential Model of Emotional Processing presented with language, imagery and content that engages men.

Using a randomized clinical trials design, this pilot project will compare the effects of the virtual intervention with a virtual control task on emotional well-being outcomes in college students.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* college student

Exclusion Criteria:

* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Patient Health Questionnaire-2 (PHQ-2) scores to 6wks post intervention | From enrollment to the end of the ~6wk follow up period.
  The scale ranges from 0-6 where higher scores indicate more dysfunction.

SECONDARY OUTCOMES:
Change from baseline Generalized Anxiety Disorder-2 scores to 6wks post intervention | From enrollment to the end of the ~6wk follow up period.
  The scale ranges from 0-6 where higher scores indicate more dysfunction.
Change from baseline Connor-Davidson Resilience Scale-2 scores to 6wks post intervention | From enrollment to the end of the ~6wk follow up period.
  Possible scores range from 0-10 where higher scores indicate higher resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Boise State University, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No